CLINICAL TRIAL: NCT00642980
Title: Randomized Multicenter Trial for the Prevention of Preterm Delivery by Testing for and Treatment of Bacterial Vaginosis in the First Trimester of Pregnancy
Brief Title: Prevention of Very Preterm Delivery by Testing for and Treatment of Bacterial Vaginosis
Acronym: PREMEVA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 060216; PHRC 2004/1918 (Other: DHOS); PHRC 2008/1929 (Other: DHOS); 2004/0428 (Other: sponsor)
Record Dates: First submitted 2008-03-21; First posted 2008-03-25 (Estimated); Last update posted 2025-10-01 (Actual); Status verified 2008-01

CONDITIONS: Pregnancy
Keywords: Pregnancy; Preterm delivery; Bacterial vaginosis; Randomized Clinical Trial; Clindamycin
MeSH Terms: conditions — Premature Birth; Vaginosis, Bacterial | interventions — Clindamycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Clindamycin Cure 1 (Active Comparator): Arm 1
  Interventions: Drug: Clindamycin
- Clindamycin Cure 2 (Active Comparator): Arm 2
  Interventions: Drug: Clindamycin
- Placebo (Placebo Comparator): Arm placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clindamycin — 300 mg capsules (per os) Intervention= 2 capsules/d during 4 days: three times a month apart
  Other Names: non applicable
  Arms: Clindamycin Cure 1
Drug: Placebo — Double blinded capsules(per os) Intervention= 2 capsules/d during 4 days: three times a month apart
  Other Names: non applicable
  Arms: Placebo
Drug: Clindamycin — 300 mg capsules (per os) Intervention= 2 capsules/d during 4 days: one time and then, after one month placebo capsules 2 capsules/d during 4 days: two times a month apart
  Other Names: non applicable
  Arms: Clindamycin Cure 2

SUMMARY:
Background. Anomalies of the vaginal flora (bacterial vaginosis, BV) are associated with an increased risk of late abortions and preterm birth. Studies of antibiotic treatment of BV to reduce the risk of prematurity have not found a statistically significant diminution of risk (<= 32 wks: OR=0.49 [0.05-5.1], < 37 wks: OR=0.83 [0.59-1.17]).A partial explanation of these findings is that some of these treatment were administered vaginally, most often during the second or third trimester

Aim: To reduce the frequency of late abortions and very preterm birth by prescribing clindamycin vs placebo to patients diagnosed with BV before 13 weeks.

DETAILED DESCRIPTION:
Patients diagnosed with BV before 13 weeks will be divided into two groups. They will be defined as at low risk when they have no history of spontaneous preterm delivery or late abortion. Women with such histories will be defined as at high risk.

Low risk patients will be asked to participate in a trial with 3 equal parallel groups, comparing two regimes of clindamycin (one or three 4-day treatments of clindamycin 300 mgx2/d) and placebo.

High-risk patients will be asked to participate in a trial with 2 parallel groups to assess the usefulness of repeating antibiotic treatment monthly by comparing the administration of one 4-day treatment of clindamycin (300 mgx2/d) to three 4-day treatments, one month apart.

ELIGIBILITY:
Inclusion Criteria:

* Nugent score >= 7
* pregnant women < 15 weeks (strictly)
* signed informed consent
* >=18 old
* speaking and understanding French language

Exclusion Criteria:

* metrorrhagias during 7 days before
* birth anticipated in an other area
* clindamycin allergy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3105 (Actual)
Dates: Start 2006-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Premature delivery (16 to 32 weeks of gestation) | At delivery

SECONDARY OUTCOMES:
Preterm labor, PPROM, Spontaneous preterm labor, PROM, Abruptio placentae, Chorioamnionitis, Fever > 38°C during labor, Post partum fever (> 38°), Post-partum wound infections, Perinatal death, NICU transfer, Bacterial neonatal colonisation. | At delivery

CONTACTS AND LOCATIONS:
Overall Officials: Damien SUBTIL, MD PhD, Principal Investigator — University Hospital, Lille (France); Gilles Brabant, MD, Study Chair — Groupe Hospitalier de l' Institut Catholique, Lille
Locations (1):
- Hopital Jeanne de Flandre, Lille, France

REFERENCES:
- [Background] Subtil D, Brabant G, Tilloy E, Devos P, Canis F, Fruchart A, Bissinger MC, Dugimont JC, Nolf C, Hacot C, Gautier S, Chantrel J, Jousse M, Desseauve D, Plennevaux JL, Delaeter C, Deghilage S, Personne A, Joyez E, Guinard E, Kipnis E, Faure K, Grandbastien B, Ancel PY, Goffinet F, Dessein R. Early clindamycin for bacterial vaginosis in pregnancy (PREMEVA): a multicentre, double-blind, randomised controlled trial. Lancet. 2018 Nov 17;392(10160):2171-2179. doi: 10.1016/S0140-6736(18)31617-9. Epub 2018 Oct 12. PMID 30322724
- See also: Website of the study (for patients and all kinds of public) — http://www.premeva.com